CLINICAL TRIAL: NCT06452784
Title: Assessment of Pre- and Postoperative Apnea-Hypopnea Index After Same-Day Discharge Bariatric Surgery in Patients With Potentially Undiagnosed Obstructive Sleep Apnea
Brief Title: Pre- and Postoperative Apnea-Hypopnea Index After Same-Day Discharge Bariatric Surgery
Acronym: DAGBAR
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-2418
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea; Bariatric Surgery Candidate; Same-day Discharge
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All study participants: Alle study participants will receive standard of care. For this study participants will complete two short questionnaires (the STOPBANG and ESS) and will undergo three home sleep apnea tests with the WatchPat one. These will be performed during the night seven days prior to surgery and during night one and three after surgery.

SUMMARY:
A recent development is same-day discharge in bariatric surgery, this seems to be safe if proper discharge criteria are used. However, yet there is no guideline for these discharge criteria, including for patients with (potential) Obstructive Sleep Apnea (OSA). To establish proper discharge criteria concerning OSA more information about (changes in) OSA during the first days after bariatric surgery is required.

The aim of this study is to assess postoperative Apnea-Hypopnea Index (AHI) changes during the first and third night after Same-Day Discharge bariatric surgery in patients with potentially untreated OSA.

Methods: Patients (n=60) will undergo a Home Sleep Apnea test , pre-operatively and during the first en third postoperative night after bariatric surgery to asses the AHI and sleep architecture.

DETAILED DESCRIPTION:
Rationale:

Bariatric surgery is a highly effective and sustainable treatment against obesity. Recently there has been a trend towards Same-Day Discharge (SDD) bariatric surgery. SDD bariatric surgery has proven to be safe, when proper discharge criteria are used. However, there is no consensus or guideline for discharge criteria for SDD bariatric surgery. In particular, discharge criteria for patients with obstructive sleep apnea (OSA) diverge between hospitals. In some, but not all hospitals, having (untreated) OSA is a contra-indication for SDD bariatric surgery.

In Rijnstate hospital, bariatric patients are not routinely tested for OSA preoperatively, meaning that they potentially have undiagnosed OSA. Having potentially undiagnosed OSA, is not a contra-indication for SDD bariatric surgery in Rijnstate hospital. Hospitals could be hesitant for SDD bariatric surgery in patients with OSA, because it is known that the apnea hypopnea index (AHI) increases postoperatively. In a population without obesity, the highest postoperative AHI was found during the third postoperative night. During this third postoperative night, patients with a normal postoperative course will already sleep at home, both after inpatient and SDD bariatric surgery. This raises the question whether having (untreated) OSA should be a contra-indication for SDD bariatric surgery. However, it is unknown if the same postoperative changes in AHI and sleep architecture occur in patients undergoing bariatric surgery. Objective: The primary objective of this study is to assess postoperative Apnea-Hypopnea Index (AHI) changes during the first and third night after Same-Day Discharge bariatric surgery in patients with potentially untreated OSA. The secondary objective of this study is to compare postoperative AHI changes between patients with a pre-operative AHI of 0-14 or ≥15. The tertiary objective of this study is to describe and compare pre- and postoperative sleep architecture.

Study design:

This is a prospective observational study. AHI and sleep architecture will be assessed and compared before and after Same-Day discharge (SDD) bariatric surgery during the first and third postoperative night with Home Sleep Apnea Tests.

Study population: Patients scheduled for primary SDD bariatric surgery without treated OSA

Main study parameters/endpoints: Primary endpoint is AHI. Secondary and tertiary endpoints are 30 days complications rate, and parameters for sleep architecture and sleep related breathing.

ELIGIBILITY:
Inclusion Criteria:

* Undergo primary bariatric surgery (Roux and y gastric bypass or sleeve gastrectomy)
* Eligible for same-day discharge
* In possession and able to use a smartphone

Exclusion Criteria:

* Revisional bariatric surgery (e.g. sleeve conversion, RYGB after gastric banding)
* Not eligible for same-day discharge
* Diagnosed OSA with treatment (CPAP, oral appliances)
* Professional drivers
* Use of alpha blockers
* Unable to speak or read the Dutch language
* Not in possession or not able to use a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary same-day discharge bariatric surgery, with exclusion of patients with treated OSA, patients using alpha blockers or professional drivers
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index (AHI) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The AHI will be measured by the Watchpat One and compared between the different timepoints.

SECONDARY OUTCOMES:
Oxygen Desaturation Index (ODI) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The ODI will be measured by the Watchpat One and compared between the different timepoints.
The AHI during rapid eye movement (sleep) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The AHI during REM sleep will be measured by the Watchpat One and compared between the different timepoints.
Respiratory disturbance index (RDI), | Measurements will take place 7 days before and 1 and 3 days after surgery
  The RDI will be measured by the Watchpat One and compared between the different timepoints.
Percentage of time with a saturation <90% | Measurements will take place 7 days before and 1 and 3 days after surgery
  The percentage of time with a saturation <90% will be measured by the Watchpat One and compared between the different timepoints.
Time of a saturation <90% | Measurements will take place 7 days before and 1 and 3 days after surgery
  Time of a saturation <90% will be measured by the Watchpat One and compared between the different timepoints.
Mean saturation | Measurements will take place 7 days before and 1 and 3 days after surgery
  Mean saturation will be measured by the Watchpat One and compared between the different timepoints.
Mean saturation during desaturations | Measurements will take place 7 days before and 1 and 3 days after surgery
  Mean desaturation during desaturations will be measured by the Watchpat One and compared between the different timepoints.
Number of desaturations | 10 days
  The number of desaturations will be measured by the Watchpat One and compared between the different timepoints.
Total sleep time (minutes) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The total sleep time will be measured by the Watchpat One and compared between the different timepoints.
Percentage of total sleep in REM sleep | Measurements will take place 7 days before and 1 and 3 days after surgery
  The percentage of REM sleep will be measured by the Watchpat One and compared between the different timepoints.
Time in REM sleep (minutes) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The time in REM sleep will be measured by the Watchpat One and compared between the different timepoints.
Percentage of total sleep in deep sleep | Measurements will take place 7 days before and 1 and 3 days after surgery
  The percentage of deep sleep will be measured by the Watchpat One and compared between the different timepoints.
The time in deep sleep (minutes) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The time in deep sleep will be measured by the Watchpat One and compared between the different timepoints.
Percentage of total sleep in light sleep | Measurements will take place 7 days before and 1 and 3 days after surgery
  The percentage of light sleep will be measured by the Watchpat One and compared between the different timepoints.
The time in light sleep (minutes) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The time in light sleep will be measured by the Watchpat One and compared between the different timepoints.
Percentage of awake time | Measurements will take place 7 days before and 1 and 3 days after surgery
  The percentage of awake time will be measured by the Watchpat One and compared between the different timepoints.
The awake time (minutes) | Measurements will take place 7 days before and 1 and 3 days after surgery
  The awake time will be measured by the Watchpat One and compared between the different timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hazebroek, Professor, Principal Investigator — Vitalys part of Rijnstate
Locations (1):
- Vitalys, Elst, Netherlands

IPD SHARING:
Plan to Share IPD: No